CLINICAL TRIAL: NCT00630981
Title: The Interest of a Specific Combined Treatment (Psychotherapy and Pharmacotherapy) in Patients With Dissociative Disorders
Brief Title: Psychotherapy and Pharmacotherapy in Dissociative Disorders
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Espace Hogan (Other)
Responsible Party: Nick Miller MD, Espace Hogan
Other Study IDs: 07-111/Psy 07-016; 07-111/Psy 07-016
Record Dates: First submitted 2008-02-28; First posted 2008-03-07 (Estimated); Last update posted 2009-04-20 (Estimated); Status verified 2009-04

CONDITIONS: Dissociative Disorders
Keywords: dissociative disorders
MeSH Terms: conditions — Dissociative Disorders | interventions — Psychotherapy; Drug Therapy; Quetiapine Fumarate; Escitalopram; Dexetimide

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Intervention group: Combined psychotherapy and pharmacological treatment
  Open single arm 'pilot' clinical trial in patients with dissociative disorders, admitted to the psychiatric emergency unit of Geneva and in the Hogan Psychotherapeutic Center in Montreux.
  Patients will be interviewed according to the Dissociative Experiences Scale (DES) and, if their score is 30 or higher, the Structured Clinical Interview for DSM-IV Dissociative Disorders (SCID) will be administered.
  Interventions: Behavioral: Psychotherapy; Drug: Pharmacological treatment (Quetiapine and/or Escitalopram)

INTERVENTIONS:
Behavioral: Psychotherapy — Specific psychotherapy for dissociative disorders
  Other Names: Dissociative Disorders
Drug: Pharmacological treatment (Quetiapine and/or Escitalopram) — Quetiapine for psychotic symptoms/Escitalopram if depressive disorders
  Other Names: Seroquel; Ketipinor; Lexapro; Cipralex

SUMMARY:
The purpose of this observational study is to measure the efficacy of a specific combined treatment (psychotherapy and pharmacotherapy) on patients with dissociative disorders, in terms of patients with a favorable outcome by means of the Dissociative Experiences Scale (DES).

DETAILED DESCRIPTION:
1. INTRODUCTION

   1. Background: Dissociative Disorders are frequent, but poorly understood and under-diagnosed [Foote et al., 2006; Spiegel, 2006], especially in psychiatric emergency units [Lazignac et al., 2005]. The management of this is commonly mixed up with psychotic, depressive and anxiety disorders.

      The treatment of the dissociative disorders remains controversial. The psychotherapeutic guidelines proposed by International Society for the Study of Dissociative Disorders (ISSD) were recently adapted for the French speaking users [Damsa et al., 2005]. There is no consensus on which antipsychotic or antidepressant would be preferable for those patients who suffer from dissociative disorders, accompanied by depressive or psychotic symptoms. We have a very good clinical experience with quetiapine and escitalopram for this specific group of patients.
   2. Rationale for this study; Clinical [Lazignac et al., 2005] and neurobiological [Kelley-Puskas et al., 2005] reviews on dissociative disorders emphasize the value of a first open label study on the effects of specific combined psychotherapy and pharmacotherapy in patients with dissociative disorders [Damsa et al., 2006].
2. STUDY OBJECTIVES

   1. Primary objective

      * The efficacy of specific combined psychotherapy and pharmacotherapy in patients with dissociative disorders, in terms of favorable outcome (DES scale).
   2. Secondary objectives

      * The efficacy of specific combined psychotherapy and pharmacotherapy in patients with dissociative disorders, in terms of DES and CGI-I scales values.
      * The effects of the combined treatment on depressive features [Hamilton Depression Rating Scale (HDRS) and the Montgomery and Asberg Depression Rating Scale items for suicide (MADRS)].
      * The occurrence of possible extra-pyramidal side effects (Barnes Akathisia and the Simpson and Angus Rating Scales).
      * The therapeutic alliance and clinical outcome (Helping Alliance Questionnaire of Luborsky), [Luborsky, 1976; Luborsky et al., 1996].
      * The relationship between serum lipid levels and depressive symptoms.
      * Tolerability and adverse effects of the quetiapine.
3. STUDY PLAN AND PROCEDURES

   1. Study design. Open single arm 'pilot' clinical trial in patients with dissociative disorders, admitted to the psychiatric emergency unit of Geneva (general capacity: 20-30 patients/day). Patients will be interviewed according to Dissociative Experiences Scale (DES) and, if their score is 30 or higher, the Structured Clinical Interview for DSM-IV Dissociative Disorders (SCID) will be administered. When the outcome on the SCID is positive, the patient can be included in the study. The Clinical Global Impression Improvement Scale (CGI-I), HDRS and the MADRS items for suicide will be administered at entry and after 3 and 8 weeks.

      The patients will be treated by a psychiatrist who has experience with the use of the specific combined treatment for dissociative disorders [Damsa et al., 2005]. The psychiatrist decides on the antidepressant/antipsychotic medication. In our unit the first choice for this indication is quetiapine (400 mg/d) for antipsychotic treatment, and escitalopram (10 mg/d) as antidepressant. The quetiapine schedule is 50-100-200-300-400-600 mg/d (min. 300 mg), then 300-600 mg/d.

      Therapeutic alliance will be assessed, both by the patient and the therapist (Luborsky scales) at the end of the first interview, and at 3 and 8 weeks. Serum lipids levels will be measured in blood samples [Agargun et al., 2004].
   2. Selection of study population

      * Inclusion criteria: written informed consent, DES-score greater than 30 and DSM-IV criteria for dissociative disorder (SCID), 18-65 years, able to comply with the study requirements, good physical health (medical history and physical examination). Female patients of childbearing potential must have a negative urinary pregnancy test.
      * Exclusion criteria: pregnancy/lactation, suicidal behavior requiring hospitalization or borderline personality disorder, substance dependence, psychotropic or cholesterol-lowering medication, intolerance or lack of response to the study medication, unstable or inadequately treated medical illness (angina pectoris, hypertension, congestive heart failure), involvement in the planning and conduct of the study, participation in the present study or in another drug trial within 4 weeks prior enrolment in study or longer in accordance with local requirements, cytochrome P450 3A4 inhibitors and inducers, absolute neutrophil count (ANC) equal or less than 1.5 x 109/L, unstable Diabetes Mellitus (DM) or opposition of physician responsible for patient's DM.
   3. Discontinuation of subjects from participation

      * Criteria: subject free withdrawal at any time, safety reasons, severe non-compliance to protocol, subject lost to follow-up, development or discover of exclusion criteria, neutrophil count of less than 1.0 x 109/L [Adverse Event (AE) specially assessed].
      * Procedures: subjects who discontinue will be asked on reason for discontinuation. If possible, they should be assessed by investigator. The investigational medication will be returned by the subject.
   4. Treatments

      * Identity of investigational product
      * Doses and treatment regimens quetiapine will be used, only if patients need an antipsychotic. Escitalopram (10 mg/day) will be used, only if patients need an antidepressant.

   Labeling of medication is in local language and complies with local regulatory requirements.

   The administration of investigational and other medication must be recorded the appropriately.
4. OUTCOME VARIABLES

   1. Primary Variable: Proportion of patients experiencing 20% DES score reduction at 8 weeks.
   2. Secondary Variables:

      * Change in DES score at 3 and 8 weeks.
      * Dichotomized DES score (into less than 25 and equal or greater than 25)
      * CGI-I score at 3 and 8 weeks
      * Barnes Akathisia and Simpson-Angus Rating Scales, Helping Alliance Questionnaire of Luborsky, Hamilton Depression Rating Scale (HDRS) and Montgomery-Asberg Depression Rating Scale items for suicide (from baseline to 3 and 8 weeks)
      * Cortisol and Lipids
      * Adverse Events
   3. Derived Efficacy Variables:

      * Favorable outcome (at least 20% reduction of DES scores).
      * Partial remission (at least 15% reduction of CGI scores).
   4. Safety measurements and variables: Cardiac frequency and blood pressure.
5. DATA MANAGEMENT. The data will be confidentially treated and will be kept in a locked room.
6. STATISTICAL METHODS AND SAMPLE SIZE

   1. Description of analysis populations:

      * The safety population consists of all patients who have taken at least one quetiapine dose.
      * The intention-to-treat (ITT) population consists of all patients who have taken at least one quetiapine dose and who have at least one baseline assessment and one post-baseline DES assessment.
      * The Per-Protocol (PP) population is a subset of the ITT population, and consists of patients who have no major protocol violations or deviations.
      * Each patient will represent one observation.
   2. Statistical analysis:

      * The primary variable: proportion of patients who experience at least 20% DES score reduction at 8 weeks for 95 % confidence interval.
      * the change in DES score, in SAS, BARS, HAM-D and Luborsky scales and in CGI-I will be analyzed by a model of analysis of covariance (ANCOVA).
      * Changes in MADRS suicidal items scores will be illustrated by descriptive statistics.
      * The relationship between therapeutic alliance and clinical outcome and between serum lipid levels and suicidal behavior will be analyzed by repeated measures ANOVA.
      * The DES score will be dichotomized into less than 25 and equal or greater than 25 and presented in frequency tables for each visit.
      * Changes in physical examination values and laboratory values will be shown in shift tables.
      * Adverse events will be summarized and shown in frequency tables.
   3. Determination of sample size: As this is a single-arm, open labeled pilot study, no formal sample size calculation is performed. In the expected sample size of 30 patients, for the proportion of patients achieving a 20% reduction in DES score, the confidence interval can be estimated between -18 and +18%; the drop-out patients will be replaced.
7. ETHICS The study protocol, including the Informed Consent Form, was approved by the local IRB Ethical committee and by the Swiss Medic Authority.

   The principal investigator is responsible for informing the IRB or IEC of any amendment to the protocol in accordance with local requirements.

   The study will be performed in accordance with ethical principles of the Declaration of Helsinki and are consistent with ICH/Good Clinical Practice, and with local regulatory requirements.

   Informed consent: The principal investigator at each centre will ensure that the subject is given full and adequate oral and written information about the nature, purpose, possible risk and benefit of the study. Subjects must also be notified that they are free to discontinue from the study at any time. The subject should be given the opportunity to ask questions and allowed time to consider the information provided.

   No study specific procedures or investigations will be performed before the subject has signed and dated the informed consent.

   The principal investigator(s) will store the original, signed Informed Consent Form. A copy of the signed Informed Consent Form will be given to the subject.
8. QUALITY CONTROL AND QUALITY ASSURANCE The study will be monitored by a designated monitor and the investigator will permit trial related audits, IRB/IEC review and regulatory inspection(s). The investigator will provide direct access to source data/documents for all quality control activities.
9. PUBLICATION POLICY Two months after study completion, abstracts for congresses and presentations will be available. Four months after study completion, a first draft of the manuscript will be available.
10. FINANCING AND INSURANCE Partial financed by AstraZeneca Insurance: Zürich Versicherung
11. PROCEDURES IN CASE OF EMERGENCY, OVERDOSE OR PREGNANCY Procedures in case of medical emergency: The principal investigator is responsible for ensuring that procedures and expertise are available to handle medical emergencies during the study. A medical emergency usually constitutes a SAE and should be reported as such, see Section 4.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written informed consent
2. DES-score greater than 30 and positive (DSM-IV) criteria for dissociative disorder using SCID for DSM IV
3. Age 18 - 65 years
4. Female patients of childbearing potential must have a negative urinary pregnancy test
5. Able to understand and comply with the requirements of the study
6. Good physical health as determined by medical history and physical examination.

Exclusion Criteria:

1. Pregnancy/lactation
2. Suicidal behaviour requiring hospitalisation or borderline personality disorder
3. Substance dependence
4. Treatment with psychotropic or cholesterol-lowering medication
5. Known intolerance or lack of response to the medication that will be prescribed in the study.
6. Unstable or inadequately treated medical illness (e.g. angina pectoris, hypertension, congestive heart failure) as judged by the investigator
7. Involvement in the planning and conduct of the study
8. Previous enrolment or randomisation of treatment in the present study.
9. Participation in another drug trial within 4 weeks prior enrolment into this study or longer in accordance with local requirements
10. The cytochrome P450 3A4 inhibitors and inducers
11. A patient with Diabetes Mellitus (DM) fulfilling one of the following criteria:

    * Unstable DM defined as enrollment glycosylated hemoglobin (HbA1c) >8.5%.
    * Admitted to hospital for treatment of DM or DM related illness in past 12 weeks.
    * Not under physician care for DM
    * Physician responsible for patient's DM care has not indicated that patient's DM is controlled.
    * Physician responsible for patient's DM care has not approved patient's participation in the study
    * Has not been on the same dose of oral hypoglycaemic drug(s) and/or diet for the 4 weeks prior to randomization. For thiazolidinediones (glitazones) this period should not be less than 8 Weeks.
    * Taking insulin whose daily dose on one occasion in the past 4 weeks has been more than 10% above or below their mean dose in the preceding 4 weeks *Note: If a diabetic patient meets one of these criteria, the patient is to be excluded even if the treating physician believes that the patient is stable and can participate in the study.
12. An absolute neutrophil count (ANC) of greater than 1.5 x 109/L

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This will be an open single arm "pilot" clinical trial on patients with dissociative disorders, admitted to the psychiatric emergency unit of Geneva and in the Hogan Psychotherapeutic Center in Montreux. Patients will be interviewed according to the Dissociative Experiences Scale (DES) and, if their score is 30 or higher, the Structured Clinical Interview for DSM-IV Dissociative Disorders (SCID) will be administered and, if the outcome on SCID is positive, the patient can be included in the study.
  The patients will be treated by a psychiatrist who has experience with the use of the specific combined treatment for dissociative disorders (Damsa et al., 2005).
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2008-02; Primary Completion 2009-04 (Actual); Study Completion 2009-07 (Estimated)

PRIMARY OUTCOMES:
To study the efficacy of a specific combined treatment (psychotherapy and pharmacotherapy) on patients with dissociative disorders, in terms of patients with a favorable outcome by means of the DES scale. | 8 weeks

SECONDARY OUTCOMES:
The relationship between serum lipid levels and depressive symptoms in patients with dissociative disorder during combined treatment. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Cristian Damsa, MD, Principal Investigator — HUG
Locations (1):
- HUG, Geneva, Canton of Geneva, Switzerland

REFERENCES:
- [Background] Agargun MY, Ozer OA, Kara H, Sekeroglu R, Selvi Y, Eryonucu B. Serum lipid levels in patients with dissociative disorder. Am J Psychiatry. 2004 Nov;161(11):2121-3. doi: 10.1176/appi.ajp.161.11.2121. PMID 15514416
- [Background] Damsa C, Pirrotta R, Adam E, Hyams H, Lazignac C, Ducrocq F. Approche thérapeutique des troubles dissociatifs. Annales Médico-Psycholgiques 163(10):902-908, 2005.
- [Background] Damsa C, Lazignac C, Pirrotta R, Andreoli A. [Dissociative disorders: clinical, neurobiological and therapeutical approaches]. Rev Med Suisse. 2006 Feb 8;2(52):400-5. French. PMID 16521716
- [Background] Foote B, Smolin Y, Kaplan M, Legatt ME, Lipschitz D. Prevalence of dissociative disorders in psychiatric outpatients. Am J Psychiatry. 2006 Apr;163(4):623-9. doi: 10.1176/ajp.2006.163.4.623. PMID 16585436
- [Background] Kelley-Puskas M, Cailhol L, D'Agostino V, Chauvet I, Damsa C. Neurobiologie des troubles dissociatifs. Annales Médico-Psycholgiques 163(10):896-901, 2005.
- [Background] Lazignac C, Cicotti A, Bortoli A-L, Kelley-Puskas M, Damsa C. Des états dissociatifs vers une clinique des troubles dissociatifs. Annales Médico-Psycholgiques 163(140): 889-895, 2005.
- [Background] Luborsky L. Helping Alliances in psychotherapy: The groundwork for a study of their relationship to its outcome. In: J.L. Cleghhorn (Ed.), Successful psychotherapy. New York, Brunner/Mazel, 92-116, 1976.
- [Background] Luborsky L, Barber JP, Siqueland L, Johnson S, Najavits LM, Frank A, Daley D. The Revised Helping Alliance Questionnaire (HAq-II) : Psychometric Properties. J Psychother Pract Res. 1996 Summer;5(3):260-71. PMID 22700294
- [Background] Spiegel D. Recognizing traumatic dissociation. Am J Psychiatry. 2006 Apr;163(4):566-8. doi: 10.1176/ajp.2006.163.4.566. No abstract available. PMID 16585425